CLINICAL TRIAL: NCT04433299
Title: Back Pain - Linking Phenotype to Pain Mechanism and Outcome.
Status: Recruiting | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00136
Record Dates: First submitted 2019-09-21; First posted 2020-06-16 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: low back pain, phenotype
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample (6 ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low back pain patients: no intervention
  Interventions: Other: no intervention, observational
- controls: no intervention
  Interventions: Other: no intervention, observational

INTERVENTIONS:
Other: no intervention, observational — no intervention, observational

SUMMARY:
To investigate whether different clinical, psychophysical and neurophysiological phenotypes can be identified among low back pain patients

DETAILED DESCRIPTION:
Low back pain patients will fill in a detailed questionnaire (incl. pain drawing) about their pain. Some of them will undergo a standardized quantitative sensory testing protocol and an fMRI procedure.

ELIGIBILITY:
Inclusion Criteria:

-primary complaint: low back pain clinically not attributable to red flags

Exclusion Criteria:

* any major medical or psychiatric condition that affects pain sensitivity
* contraindications to MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 80 with low back pain
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
spatial pain extent | baseline
  spatial pain extent (body map)
measures for central sensitization | baseline
  temporal summation and conditioned pain modulation

SECONDARY OUTCOMES:
changes in spatial pain extent | changes from baseline to 3 months
  changes in spatial pain extent (bodymap)
changes in measures for central sensitization | changes from baseline to 3 months
  changes in temporal summation and conditioned pain modulation

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, MD, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sirucek L, De Schoenmacker I, Gorrell LM, Lutolf R, Langenfeld A, Baechler M, Wirth B, Hubli M, Zolch N, Schweinhardt P. The periaqueductal gray in chronic low back pain: dysregulated neurotransmitters and function. Pain. 2025 May 15;166(7):1690-1705. doi: 10.1097/j.pain.0000000000003617. PMID 40372313